CLINICAL TRIAL: NCT02300883
Title: Diagnostic and Prognostic Role of New Inflammation Biomarkers in Patients With Malignant Pleural Mesothelioma
Brief Title: Observational Prospective Analysis of Biological Characteristics of Mesothelioma Patients
Status: Completed | Type: Observational
Sponsor: Armando Santoro, MD (Other)
Responsible Party: Sponsor-Investigator, Armando Santoro, MD, Principal Investigator, Istituto Clinico Humanitas
Organization: Istituto Clinico Humanitas (Other)
Other Study IDs: ONC/OSS-02/2011
Record Dates: First submitted 2013-05-27; First posted 2014-11-25 (Estimated); Last update posted 2022-09-09 (Actual); Status verified 2022-09

CONDITIONS: Malignant Mesothelioma
MeSH Terms: conditions — Mesothelioma, Malignant

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — pleural effusion
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- no treatment: no treatment

SUMMARY:
This is an observational prospective analysis of biological characteristics of malignant mesothelioma (MM) patients. Frozen and paraffin-embedded tumor specimens and pleural effusion of patients will be collected and than will be analyzed with the following analyses:

1Purification of Tumour Associated Macrophages (TAM) and tumour cells from pleural effusions.

2.Mass spectrometry analysis of TAMs and tumor cells 3.Co focal microscopy analysis of macrophages, tumour cells and specimens derived from patients.

DETAILED DESCRIPTION:
This is an observational prospective analysis of biological characteristics of malignant pleural mesothelioma (MPM) patients. Frozen and paraffin-embedded tumor specimens and pleural effusion of patients will be collected and than will be analyzed with the following analyses:

1. Purification of TAMs and tumour cells from pleural effusions. Pleural effusions will be subjected to centrifugation in order to separate cellular and non-cellular components. Cell-free supernatant will be collected and subjected to further analysis for the identification and characterization of secreted proteins (ELISA, Western Blot). Pleural effusion cell components will be characterized by cytofluorimetry in order to evaluate leukocytes composition (e.g. macrophages, neutrophils, lymphocytes). Next, to isolate TAMs from the cellular components, the investigators will adopt a standard protocol currently performed in the investigators group to purify TAMs from ascites derived from ovarian carcinoma patients . Briefly, TAMs will be separated by their selective capacity to adhere in culture plates in serum-free conditions. After 1 hour of incubation, non-adherent cells (mainly tumour cells and other inflammatory cells) will be thoroughly washed off with jets of medium. After adherence, cells were rested for 1 hour in standard culture conditions and subsequently lysed to extract proteins. To isolate tumour cells from leukocytes, a cell sorting-based approach will be used. Briefly, inflammatory cells will be stained with lymphocyte common antigen (CD45) antibody and negative cells (tumour cells) will be separated by cell sorting. Next tumour cells will be grown and amplified in standard culture conditions.
2. Mass spectrometry analysis of TAMs and tumor cells Generation of proteome and the phospho-proteomic maps of TAMs and tumour cells will be accomplished by quantitation of both the entire proteome and the phospho-proteome. Results obtained with TAMs will be compared to untreated, M1 and M2 polarized Monocytes-derived macrophages (M-DM), while tumor cells purified from patients' pleural effusion will be analysed with respect to human mesothelial cells. Protein samples obtained from the purified TAMs and tumour cells, derived from the patient's pleural effusions, will be extracted using lysis/acetone precipitation. Cell extracts will be subsequently subjected to trypsin digestion and the resulting peptides will be labelled with the "iTRAQ" reagents. Labelled peptides will be separated with the first dimension of the separation being strong cation exchange (SCX) chromatography. Fractions will be collected and phospho-enriched, when required. The pooled mixture of peptides will be submitted to a second dimension chromatographic separation, organized as a two-step process: a desalting/concentrating pre-column, and an analytical column for the separation. System is a nano-flow configuration, with direct interfacing to a mass spectrometer. Tandem mass spectrometry will be performed on a hybrid ion-trap (IT) - Fourier transform ion-cyclotron-resonance mass spectrometer. Quantitative and identification data analysis will be carried out with Proteome Discoverer software (Thermo), using SEQUEST as the search engine. Statistical analysis and data classification will be carried out with aid of in-house written script for the freeware statistical analysis package.
3. Co focal microscopy analysis of macrophages, tumour cells and specimens derived from patients. The analysis will be conducted on the cellular components derived from pleural effusion (as previously described) and from frozen and paraffin-embedded tissues. Immunofluorescence staining will be performed with markers of DNA damage and polarized inflammation. Furthermore, immunofluorescence analysis will be held to validate putative new MM molecular markers obtained from the mass spectrometry studies.

ELIGIBILITY:
Inclusion Criteria:

* Malignant pleural mesothelioma patients
* Availability of plural effusion and frozen and paraffin-embedded tumor specimens.

Exclusion Criteria:

* Unavailability of plural effusion and frozen and paraffin-embedded tumor specimens.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Malignant pleural mesothelioma patients
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2011-04; Primary Completion 2017-12 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
dissect the molecular mechanisms underlying the development of malignant mesothelioma | 24 months
  characterization of the microenvironment (expression of M1 and M2 markers of polarized inflammation - cytokines and chemokines inducers or inhibitors of the inflammatory response) and the interplay between tumour cells and TAMs (expression of DNA damage markers) in order to dissect the molecular mechanisms underlying the development of malignant mesothelioma

SECONDARY OUTCOMES:
study of the effect of TAMs | 24 months
  the study of the effect of TAMs on the induction of the DNA damage on (Human mast cell) HMC cells, and a possible synergic effect with asbestos fibers;
investigation of molecular mechanisms linking macrophages | 24 months
  the investigation of molecular mechanisms linking macrophages polarized activation with asbestos-induced mesothelioma
molecular characterization (proteome) of TAMs and tumor cells | 24 months
  the molecular characterization (proteome) of TAMs and tumor cells, isolated from pleural effusion derived from patients
compare in specimens from mesothelioma patients and the candidate molecular markers | 24 months
  to compare in specimens from mesothelioma patients and the candidate molecular markers, obtained expression in the above-mentioned tasks
Investigate the association of selected markers with Overall Survival | 24 months
  To Investigate the association of selected markers with Overall Survival (OS)

CONTACTS AND LOCATIONS:
Overall Officials: armando Santoro, MD, Principal Investigator — Istituto Clinico Humanitas
Locations (2):
- Italy (2):
  - Istituto Clinico Humanitas, Rozzano, Milano
  - Istituto Clinico Humanitas, Rozzano, Milan

IPD SHARING:
Plan to Share IPD: No
not planned